CLINICAL TRIAL: NCT05617703
Title: Evaluation of Glass Ionomer With Advanced Glass Hybrid Technology Versus Resin Modified Glass Ionomer in Adult Patients With Carious Cervical Lesions After One Year: Randomized Clinical Trial
Brief Title: Evaluation of Glass Ionomer With Advanced Glass Hybrid Technology Versus Resin Modified Glass Ionomer in Adult Patients With Carious Cervical Lesions After One Year
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Magdy Zayed, masters degree student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14422018462089
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Dental Caries Class v
MeSH Terms: interventions — glass ionomer

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups with a 1:1 allocation using computer generated randomization list (www.random.org).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double blinded study. The participants will not be informed to which group they will be assigned. The operator will be blinded because the restorative procedures for both groups are the same, the outcome assessors will not be informed about the type of restoration they evaluate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glass Ionomer with Advanced Glass Hybrid Technology (Equia forte HT fil, GC, Japan) (Experimental): Glass Hybrid restorative systems in the clinical point of view are self-cure bulk fill materials laminated with a nano-filled, self-adhesive resin coat.
  Nowadays, a new glass hybrid innovation called Advanced Glass Hybrid technology was achieved through introduction of ultra-fine highly reactive glass and high-molecular weight polyacrylic acid powders within conventional glass using prefractive indexes.
  Interventions: Drug: Glass Ionomer with Advanced Glass Hybrid Technology (Equia forte HT fil, GC, Japan)
- Resin Modified Glass Ionomer (Fugi II LC, GC, Japan). (Active Comparator)
  Interventions: Drug: Glass Ionomer with Advanced Glass Hybrid Technology (Equia forte HT fil, GC, Japan)

INTERVENTIONS:
Drug: Glass Ionomer with Advanced Glass Hybrid Technology (Equia forte HT fil, GC, Japan) — Advanced Glass Hybrid technology (AGH) was achieved through introduction of ultra-fine highly reactive glass and high-molecular weight polyacrylic acid powders within conventional glass using particles and fillers with close refractive indexes

SUMMARY:
The goal of this [type of study: Randomized clinical trial] to compare the clinical performance of using glass ionomer with advanced glass hybrid technology (AGH) in cervical carious lesion, versus Resin modified glass ionomer (RMGI) using esthetic and mechanical properties according to FDI criteria over one year.

in adult patients with cervical carious lesion.

The main question it aims to answer are:

• Will the use of glass ionomer with advanced glass hybrid technology, achieved through introduction of ultra-fine highly reactive glass and high-molecular weight polyacrylic acid powders within conventional glass ,or Resin Modified Glass Ionomer have better mechanical and estheic properties over one year in adult patients with cervical carious lesions ?

Participants will be assessed for medical and dental histories first. Then an examination of the patients will be done using visual inspection by using a dental mirror and probe. Eligible patients according to inclusion and exclusion criteria will be informed about all procedures with follow up time if they accept, their signature on written informed consents will be obtained. Eligible participants will be randomly divided into two groups according to the type of restoration that will be received after class V cavity preparations for carious cervical lesions.

Patients will be given local anaesthesia (Mepecaine - L Cartridges) as required, and the teeth will be isolated. A No. #330 bur (MANI, INC, Japan) in a high-speed hand piece with air/water coolant will be used to prepare class V cavity. Sharp excavators of suitable size were used to excavate soft carious lesions in dentin. the prepared cavity will be isolated with rubber dam.

The first group (A) will be received resin modified glass ionomer restorative material and the second group (B) will be received advanced glass hybrid glass ionomer . Each restoration will be evaluated for clinical parameters after finishing and polishing at baseline and regular recalls of 6 months and one year. The restorations will be clinically examined according to FDI criteria criteria in terms of esthetic and mechanical properties . The information that will be obtained will be collected and statistically analyzed.

DETAILED DESCRIPTION:
Eligibility criteria

The participants were chosen according to the following eligibility criteria:

Inclusion criteria Exclusion criteria

Patient inclusion:

1. Patients aging ≥18 years.
2. Patients with High caries risk.
3. Patients with untreated cervical caries lesion that need restorative treatment.
4. Males or females
5. No abnormal occlusion for selected teeth.
6. Patients with good likelihood of recall availability

Tooth inclusion:

1. Permanent teeth.
2. Absence of mobility.
3. Primary carious lesions.
4. Vital with positive reaction to thermal stimulus .

Patient exclusion:

1. Participants with general/systemic illness.
2. Concomitant participation in another research study.
3. Inability to comply with study procedures.
4. Heavy bruxism habits.
5. Last experience with allergic reactions against any components of the used materials.
6. Patients receiving orthodontic treatment.
7. Teeth supporting removable prosthesis
8. Patients with cervical caries lesions that need crown restoration.
9. Xerostomia.

Tooth exclusion:

1. Teeth with clinical symptoms of pulpitis such as spontaneous pain or sensitivity to pressure.
2. Non-vital teeth.
3. Periapical Abscess or Fistula.

   * Outcomes:

For each recall examination, two independent evaluators will perform the direct clinical evaluation at baseline, after 6 and 12 months using written criteria based on FDI criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patient inclusion:

  1. Patients aging ≥18 years.
  2. Patients with High caries risk.
  3. Patients with untreated cervical caries lesion that need restorative treatment.
  4. Males or females
  5. No abnormal occlusion for selected teeth.
  6. Patients with good likelihood of recall availability

Tooth inclusion:

1. Permanent teeth.
2. Absence of mobility.
3. Primary carious lesions.
4. Vital with positive reaction to thermal stimulus .

Exclusion Criteria:

* 1. Participants with general/systemic illness. 2. Concomitant participation in another research study. 3. Inability to comply with study procedures. 4. Heavy bruxism habits. 5. Last experience with allergic reactions against any components of the used materials.

  6. Patients receiving orthodontic treatment. 7. Teeth supporting removable prosthesis 8. Patients with cervical caries lesions that need crown restoration. 9. Xerostomia.

Tooth exclusion:

1. Teeth with clinical symptoms of pulpitis such as spontaneous pain or sensitivity to pressure.
2. Non-vital teeth.
3. Periapcal Abscess or Fistula.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
FDI criteria | one year
  Esthetic and mechanical evaluation

IPD SHARING:
Plan to Share IPD: Yes
international and national publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code